CLINICAL TRIAL: NCT06566911
Title: A Pilot Study on AI-Based Voice Analysis for Monitoring Patients Hospitalized With Acute Decompensated Heart Failure
Brief Title: Voice Analysis for Monitoring Patients With Heart Failure
Acronym: VAMP-HF
Status: Recruiting | Type: Observational
Sponsor: Noah Labs (Industry)
Collaborators: Charite University, Berlin, Germany (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-011322
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study involves ADHF patients at two sites in the United States and Germany. After informed consent and screening assessments, participants will perform daily voice recordings during their hospital stay, from admission until discharge. Alongside voice data, additional clinical information such as left ventricular ejection fraction, NTpro-BNP levels, and ECG-data will be collected for comprehensive analysis. The study's goal is to identify voice-based indicators of heart failure progression, with the potential to enhance remote monitoring and self-management strategies for heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Acutely Decompensated Heart Failure.
* At least 18 years of age.

Exclusion criteria:

* Disabling mental diseases (e.g., Alzheimer's disease)
* Clinically diagnosed chronic obstructive pulmonary disease (COPD)
* Treatment in ICU or IMU
* Dialysis treatment
* Previous operations on organs involved in generation of voice (vocal tract, vocal folds, etc.)
* Neurodegenerative diseases
* Pregnancy
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients, aged 18 and older, hospitalized with acutely decompensated heart failure, irrespective of left ventricular ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in vocal characteristics from admission to discharge and their correlation with heart failure severity markers. | Hospital stay
  The primary endpoint is the change in vocal characteristics from admission to discharge, and its correlation with clinical markers of heart failure severity, such as weight change from admission to discharge, NTpro-BNP levels, ECG-parameters, and left ventricular ejection fraction (LVEF).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — German Heart Institute
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Deutsches Herzzentrum der Charité, Berlin, Germany